CLINICAL TRIAL: NCT00446784
Title: A Phase 1, Double Blind Study Of The Safety And Pharmacokinetics Of Multiple Doses Of CE 224,535 In Subjects With Rheumatoid Arthritis Receiving Methotrexate
Brief Title: Study Of The Safety Of CE 224,545 And Methotrexate In Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6341006
Record Dates: First submitted 2007-03-09; First posted 2007-03-13 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — CE 224,535; Methotrexate

INTERVENTIONS:
Drug: CE-224,535
Drug: Methotrexate

SUMMARY:
CE 224,535 is being developed for the treatment of rheumatoid arthritis. The purpose of this study is to evaluate the safety and tolerability of CE 224,535 after 4 weeks of treatment in subjects with rheumatoid arthritis already receiving methotrexate

ELIGIBILITY:
Inclusion Criteria:

* Adults patients with rheumatoid arthritis
* Patients who have received stable weekly doses of oral methotrexate (5 to 25 mg/week administered as a single dose) for a minimum of 28 days (4 weeks/4 doses)

Exclusion Criteria:

* History of chronic infectious disease such as genitourinary, pulmonary or sinus infections.
* Any current or known malignancy or history of malignancy within the previous 5 years
* Pregnant or lactating women; women of child-bearing potential who are unwilling to unable to use an acceptable method of birth control during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2007-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events throughout the study

SECONDARY OUTCOMES:
Pharmacokinetics of CE 224,535 on Days 7 and 8
Pharmacokinetics of Methotrexate on Days 1 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Ducansville, Pennsylvania

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6341006&StudyName=Study%20Of%20The%20Safety%20Of%20CE%20224%2C545%20And%20Methotrexate%20In%20Patients%20With%20Rheumatoid%20Arthritis